CLINICAL TRIAL: NCT05071898
Title: Pharmacogenetics of Response to GLP1R Agonists
Acronym: PORT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Amber Beitelshees, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP00097563
Record Dates: First submitted 2021-09-27; First posted 2021-10-08 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Diabetes Type 2
Keywords: GLP-1 receptor agonist; Insulin secretion; Insulin sensitivity; Pharmacogenomics; Semaglutide
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: The study will employ a paired design with each participant being studied both before and after receiving semaglutide treatment for six weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label administration of semaglutide (Experimental): Semaglutide: 0.25 mg, sc, q.week for 4 weeks followed by 0.5 mg, sc, q.week for 2 weeks
  Interventions: Drug: Semaglutide Pen Injector [Ozempic]

INTERVENTIONS:
Drug: Semaglutide Pen Injector [Ozempic] — Participants will receive subcutaneously injected semaglutide (0.25 mg/wk) for 4 weeks followed by semaglutide (0.5 mg/wk) for an additional two weeks.
  Other Names: Ozempic; Wegovy

SUMMARY:
Overweight/obese otherwise healthy volunteers will be recruited from the Old Order Amish population in Lancaster County, PA. Lancaster County, PA. Pharmacodynamic responses to GLP1R agonist will be assessed by conducting frequently sampled intravenous glucose tolerance tests (FSIGT) both before and after semaglutide for six weeks. The proposal proposes two specific aims:

1. Specific Aim #1. To identify genetic variants associated with effects of a GLP1R agonist to enhance glucose-stimulated first phase insulin secretion in the two FSIGTs (before and after administration of drug).
2. Specific Aim #2. To identify genetic variants associated with the effect of a GLP1R agonist to accelerate the rate of glucose disappearance as assessed in the two FSIGTs (before and after administration of drug).

Genotyping will be conducted using a high-density array with comprehensive coverage of DNA sequence variants. In addition, the analysis will leverage a global imputation panel generated from 1,025 Amish individuals.

DETAILED DESCRIPTION:
Overweight/obese otherwise healthy volunteers will be recruited from the Old Order Amish population in Lancaster County, PA. In order to assess pharmacodynamic responses, research participants will undergo two frequently sampled intravenous glucose tolerance tests (FSIGT). The first FSIGT will be conducted at baseline prior to administration of drug. The second FSIGT will be conducted after six weeks of treatment with semaglutide (0.25 mg/wk X 4 wks; 0.5 mg/sk X 2 wks). The proposal proposes two specific aims:

* Specific Aim #1. To identify genetic variants associated with effects of a GLP1R agonist to enhance glucose-stimulated first phase insulin secretion in the two FSIGTs (before and after administration of drug).
* Specific Aim #2. To identify genetic variants associated with the effect of a GLP1R agonist to accelerate the rate of glucose disappearance as assessed in the two FSIGTs (before and after administration of drug).

After being determined to be eligible and after having given informed consent, participants will undergo two frequently samples intravenous glucose tolerance tests conducted at two clinic visits as described below:

Visit #1 - Research participants will be transported to the Amish Research clinic in the fasting state (minimum of 8 hour, maximum of 24 hour fast) where height, weight, waist and hip measurements, and vital signs will be measured. Women of child-bearing potential will undergo a urine pregnancy test. An FSIVGTT will be conducted as follows: IV (intravenous) access will be established in both arms of the research participant, one for glucose infusion and the other for frequent blood sampling. NSS (normal saline solution) will be used to maintain patency of IV. Intravenous glucose (0.3 g/kg) will be infused over 2 min at time=0, and 31 blood samples will be obtained between -15 and +180 minutes. Approximately 180 ml (36 tsp.) of blood will be drawn. Upon completion of the FSIVGTT, the participant will be instructed in the self-administration of subcutaneous (s.c.) injection of semaglutide. The first dose of semaglutide .25mg will be administered at this time. The participant will be provided with a post-fasting meal.

Home self-administration of weekly semaglutide: The participant will self-administer s.c. semaglutide weekly for 5 weeks (.25 mg for weeks 2,3,4 and .5 mg for weeks 5,6) A research nurse may observe the participant self-administering the first home dose and will make additional home visits as needed to ensure successful self-injection. The participant will use the study provided scale to obtain and record daily weights in the morning before breakfast throughout the medication weeks.

Visit #2 - This visit will be scheduled within 1 week of the final (6th) dose of semaglutide +/- 5 days. The FSIVGTT will be conducted exactly as during the previous clinic visit.

Genotyping will be conducted using a high-density array with comprehensive coverage of DNA sequence variants. The project will leverage a global imputation panel generated from whole genome sequence data on ~ 100K subjects including 1,025 Amish individuals obtained through the NHLBI-sponsored Trans-Omics for Precision Medicine (TOPMed) program.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 27 kg/m2
* Of Amish Descent

Exclusion Criteria:

* Woman of childbearing age who is sexually active
* History of diabetes (HbA1c > 6.5% or random glucose >200 mg/dL)
* Known allergy to semaglutide
* Medical issues, which in the judgment of the research physician or PIs might increase the risk associated with participation in the study
* eGFR < 60 mL/min/1.73 sq. m.
* Hematocrit < 35%
* TSH < 0.4 o4 > 5.5
* AST or ALT in excess of 2X the upper limit of normal
* Unable to discontinue a drug, vitamin, or nutritional supplement, which in the judgment of the research physician or PIs might alter the response to semaglutide
* Personal or family history of medullary carcinoma of the thyroid or multiple endocrine neoplasia, type 2

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals will self-identify as being male, female, or other non-binary gender identity. Although we anticipate that most Amish will self-identify as being either male or female, everyone is potentially eligible regardless of their gender identity.
Enrollment: 600 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
First phase insulin secretion | Measured both at baseline and after completing 6 weeks of semaglutide therapy
  Area under the curve for plasma insulin levels measured at times between 0-10 min after administration of intravenous glucose (0.3 g/kg)
Second phase insulin secretion | Measured both at baseline and after completing 6 weeks of semaglutide therapy
  Area under the curve for plasma insulin levels measured at times between 10-50 min after administration of intravenous glucose (0.3 g/kg)
Rate of glucose disappearance | Measured both at baseline and after completing 6 weeks of semaglutide therapy
  Slope of the plot of log(glucose concentration) as a function of time. This will be calculated based on a linear regression using data points between 25-50 minutes after administration of intravenous glucose (0.3 g/kg)

SECONDARY OUTCOMES:
Weight loss | Assessed after completing 6 weeks of semaglutide therapy
  This will be measured as the baseline weight in kg minus the weight after completing 6 weeks of semaglutide therapy.

OTHER OUTCOMES:
Insulin sensitivity (Si) | Measured both at baseline and after completing 6 weeks of semaglutide therapy
  Estimated using Bergman's minimal model
Glucose effectiveness (Sg) | Measured both at baseline and after completing 6 weeks of semaglutide therapy
  Estimated using Bergman's minimal model

CONTACTS AND LOCATIONS:
Overall Officials: Amber L Beitelshees, PharmD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Amish Research Clinic, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Within the constraints of assuring confidentiality of research participants, we plan to share deidentified IPD within two years after the study investigators have published the results of the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Two years after PIs have published the results of the clinical trial
Access Criteria: Academic researchers who sign data sharing agreement to protect the confidentiality of the participants.

REFERENCES:
- [Derived] Taylor SI, Montasser ME, Yuen AH, Fan H, Yazdi ZS, Whitlatch HB, Mitchell BD, Shuldiner AR, Muniyappa R, Streeten EA, Beitelshees AL. Acute pharmacodynamic responses to exenatide: Drug-induced increases in insulin secretion and glucose effectiveness. Diabetes Obes Metab. 2023 Sep;25(9):2586-2594. doi: 10.1111/dom.15143. Epub 2023 Jun 1. PMID 37264484